CLINICAL TRIAL: NCT03927638
Title: Differences in Sitting Versus Standing on Metabolic and Cardiovascular Measurements
Status: Enrolling by invitation | Type: Observational
Sponsor: Montclair State University (Other)
Responsible Party: Principal Investigator, Peter A. Hosick, Assistant Professor, Montclair State University
Other Study IDs: 17-18-861
Record Dates: First submitted 2019-04-22; First posted 2019-04-25 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2024-10

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Normal Weight: Group is determined based upon subjects weight status. Subjects will preform computer work in the seated and standing position in a counterbalanced manner while metabolic and cardiovascular measurements are made.
  Interventions: Behavioral: sit/stand
- Overweight/Obese: Group is determined based upon subjects weight status. Subjects will preform computer work in the seated and standing position in a counterbalanced manner while metabolic and cardiovascular measurements are made.
  Interventions: Behavioral: sit/stand

INTERVENTIONS:
Behavioral: sit/stand — Subjects will be asked to both sit and stand during a single trial.

SUMMARY:
This investigations examined the effect that posture has on metabolic and cardiovascular measurements. Further, it will explore the potential for body weight status or physical activity to influence these relationships. All subjects will complete a seated condition and a standing condition in a counterbalanced manner.

DETAILED DESCRIPTION:
The purpose of the present study was to evaluate both metabolic and cardiovascular responses to acute bouts of computer work while sitting and standing. Cardiovascular measurements were made using continuous non-invasive blood pressure monitoring and metabolic measurements were made using indirect calorimetry. Subjects will be grouped and analyzed based upon the weight status of the subject. All subjects will complete a seated condition and a standing condition in a counterbalanced manner. Investigators hypothesize that metabolic and cardiovascular responses will be elevated in the standing condition compared to sitting.

ELIGIBILITY:
Inclusion Criteria:

* healthy adult

Exclusion Criteria:

* Have a history of cancer, cardiac issues, hypertension, pulmonary disease, stroke, neurological or muscular dystrophy, uncontrolled diabetes, or any life threatening chronic conditions.
* Are currently being treated for infectious mononucleosis, hepatitis, pneumonia, or other infectious diseases.
* Are unable or unwilling to stand in one position continuously for 15-20 minutes at a time.
* Use nicotine products, or non-contraceptive hormonal therapy (birth control is okay).
* Are pregnant or trying to become pregnant.
* Are not between 18 and 50 years of age.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Healthy subjects between the ages of 18 and 50 years.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2018-11-11 (Actual); Primary Completion 2028-05-15 (Estimated); Study Completion 2028-05-15 (Estimated)

PRIMARY OUTCOMES:
Heart Rate | Approximately 15 minutes in each condition (sitting and standing)
  Using human non-invasive blood pressure continuous monitoring placed on the middle finger of the non-dominant hand will be used to measure heart rate based upon beat-by-beat finger pressure.
Systolic Blood Pressure (SBP) | Approximately 15 minutes in each condition (sitting and standing)
  Using human non-invasive blood pressure continuous monitoring placed on the middle finger of the non-dominant hand will be used to measure SBP based upon beat-by-beat finger pressure.
Diastolic Blood Pressure (DBP) | Approximately 15 minutes in each condition (sitting and standing)
  Using human non-invasive blood pressure continuous monitoring placed on the middle finger of the non-dominant hand will be used to measure DBP based upon beat-by-beat finger pressure.
Oxygen Consumption | Approximately 15 minutes in each condition (sitting and standing)
  Oxygen consumption will be measured using indirect calorimetry.
Carbon Dioxide Production | Approximately 15 minutes in each condition (sitting and standing)
  Carbon Dioxide will be measured using indirect calorimetry.
Ventilation | Approximately 15 minutes in each condition (sitting and standing)
  Ventilation will be measured using indirect calorimetry.
Respiratory Exchange Ration (RER) | Approximately 15 minutes in each condition (sitting and standing)
  RER will be calculated using oxygen and carbon dioxide value measure from indirect calorimetry.

SECONDARY OUTCOMES:
Height | 1 minute
  Standard stadiometer will be used to measure height in meters.
Weight | 1 minute
  Standard scale will be used to measure weight in kilograms.
Body Mass Index (BMI) | 1 minute
  Height in meters and weight in kilograms will be used to calculate BMI using the formula BMI = kg/m^2.
Body Composition | Approximately 15 minutes
  Body composition will be measured using air displacement plethysmography.
Total Peripheral Resistance (TPR) | Approximately 15 minutes in each condition (sitting and standing)
  Using human non-invasive blood pressure continuous monitoring placed on the middle finger of the non-dominant hand will be uses to estimate TPR based upon beat-by-beat finger pressure.
Stroke Volume | Approximately 15 minutes in each condition (sitting and standing)
  Using human non-invasive blood pressure continuous monitoring placed on the middle finger of the non-dominant hand will be used to estimate TPR based upon beat-by-beat finger pressure.
Cardiac Output (Q) | Approximately 15 minutes in each condition (sitting and standing)
  Using human non-invasive blood pressure continuous monitoring placed on the middle finger of the non-dominant hand will be used to estimate Q based upon beat-by-beat finger pressure.
Muscle Oxygen Saturation | Approximately 15 minutes in each condition (sitting and standing)
  Using Near-inferred spectroscopy muscle oxygen consumption will be monitored.

CONTACTS AND LOCATIONS:
Locations (1):
- Montclair State University, Montclair, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hosick PA, Willett JM, Matthews EL. Cardiovascular strain and metabolic rate are higher following 15 minutes of standing versus seated computer work. Eur J Prev Cardiol. 2020 Dec;27(19):2131-2133. doi: 10.1177/2047487319867402. Epub 2019 Jul 29. No abstract available. PMID 31357884